CLINICAL TRIAL: NCT05463016
Title: Immediate and Extended Wear Impact of Color Correcting Lenses on Color Vision Deficiency
Brief Title: Impact of Color Correcting Lenses on Color Vision Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, JEFFREY CARL RABIN, Professor, University of the Incarnate Word
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022-1194-EXP; 1T35EY032441-01A1 (NIH)
Record Dates: First submitted 2022-07-03; First posted 2022-07-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Color Blindness; Color Vision Defects; Color Blindness, Green; Color Blindness, Red
Keywords: Color-Correcting Lenses
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Intervention Model Description: Double blind randomized crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Color Vision Deficient with Color Correcting Lenses (Experimental): 10 subjects confirmed to have hereditary color vision deficiency randomly assigned to experimental group 1 which includes baseline testing with and without color correcting lenses, followed by 7 days of wear, minimum 3 hours/day, followed by retesting with and without color correcting lenses.
  Interventions: Device: Experimental Group 1: Color Correcting Lenses
- Color Vision Deficient with Placebo Lenses (Placebo Comparator): 10 subjects confirmed to have hereditary color vision deficiency randomly assigned to Placebo Group 1 which includes baseline testing with and without placebo lenses, followed by 7 days of wear, minimum 3 hours/day, followed by retesting with and without placebo lenses.
  Interventions: Device: Placebo Group 1: Placebo Lenses
- Crossover: Placebo to Experimental (Experimental): Placebo Group 1 crosses over to become Experimental Group 2 which includes baseline testing with and without color correcting lenses, followed by 7 days of wear, minimum 3 hours/day, followed by retesting with and without color correcting lenses.
  Interventions: Device: Placebo Group 1 Crosses over to become Experimental Group 2: Color Correcting Lenses
- Crossover: Experimental to Placebo (Placebo Comparator): Experimental Group 1 crosses over to become Placebo Group 2 which includes baseline testing with and without placebo lenses, followed by 7 days of wear, minimum 3 hours/day, followed by retesting with and without placebo lenses.
  Interventions: Device: Experimental Group 1 Crosses over to become Placebo Group 2: Placebo Lenses
- Control Group: Subjects with Normal Color Vision (Active Comparator): Fifteen subjects confirmed to have normal color vision will be tested in a single session to determine whether color correcting lenses affect color vision in color vision normal subjects and to provided normative data for several unique measures of color vision performance
  Interventions: Device: Color Correcting Lenses in Subjects with Normal Color Vision

INTERVENTIONS:
Device: Experimental Group 1: Color Correcting Lenses — Color Correcting Lenses
  Arms: Color Vision Deficient with Color Correcting Lenses
Device: Placebo Group 1: Placebo Lenses — Placebo Lenses
  Arms: Color Vision Deficient with Placebo Lenses
Device: Placebo Group 1 Crosses over to become Experimental Group 2: Color Correcting Lenses — Color Correcting Lenses
  Arms: Crossover: Placebo to Experimental
Device: Experimental Group 1 Crosses over to become Placebo Group 2: Placebo Lenses — Placebo Lenses
  Arms: Crossover: Experimental to Placebo
Device: Color Correcting Lenses in Subjects with Normal Color Vision — Color Correcting Lenses
  Arms: Control Group: Subjects with Normal Color Vision

SUMMARY:
To demonstrate improved color vision in subjects with color vision deficiencies while wearing color-correcting lenses and after color-correcting lense use.

DETAILED DESCRIPTION:
The long term objective of this study is to extend upon research demonstrating improvements in color vision deficiencies (CVDs) while wearing color-correcting lenses (CCLs) and after wearing CCLs. Recordings of brainwaves and eye-waves will be made to assess the retina, optic nerve and brain in order to localize where adaptive changes in the visual system are occurring in response to wearing CCLs.

ELIGIBILITY:
Inclusion Criteria:

* no reported history of eye, systemic or ocular disease
* VA of 20/30 in each eye
* hereditary color vision deficient (CVDs) verified by failing scores on the red-green anomaloscope (outside system normal range) and Ishihara testing (3 or more errors on 14 testable plates)
* color vision normal (CVNs) verified by passing red-green anomaloscope (outside system normal range) and Ishihara testing (3 or more errors on 14 testable plates)

Exclusion Criteria:

* reported use of sleep-inducing or wakefulness drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Cone Contrast Test | 2 WeekS
  Cone Contrast Sensitivity (CS) Test (CCT, Innova Systems, Inc.): red, green & blue cone CS using 100-point scale based on log changes in CS. Values will be converted to Z-scores to compare to outcomes with other units.
Cone Contrast Naming Test | 2 Weeks
  Red, green & blue cone CS and color naming accuracy each based on 100-point scale. Values will be converted to Z-scores to compare to outcomes with other units.
Letter Chart Testing | 2 Weeks
  Letter chart cone specific VA, small letter CS, and large letter CS scored as number of letters correct with VA expressed as log MAR & CS as log CS. Values will be converted to Z-scores to compare to outcomes with other units.
Color Matching | 2 Weeks
  Cone specific color matching provides the contrast seen by the normal cone type which matches the contrast seen by the defective cone type in units of % Weber contrast. Values will be converted to Z-scores to compare to outcomes with other units.
Color Identification Test | 2 Weeks
  Cockpit color identification test measure reaction time in seconds and error rate to identify colored targets on a computer display. Values will be converted to Z-scores to compare to outcomes with other units.
Visual Electrodiagnostic Testing | 2 Weeks
  Cone specific visual brainwaves (VEPs) and flash and pattern eye waves (ERGs) will be quantified in terms of amplitude in microvolts and latency in msec. Values will be converted to Z-scores to compare to outcomes with other units.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rabin, Principal Investigator — C
Locations (1):
- University of the Incarnate Word Rosenberg School of Optometry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the data with anyone outside the research team.

REFERENCES:
- [Background] Cole BL, Maddocks JD. Color vision testing by Farnsworth lantern and ability to identify approach-path signal colors. Aviat Space Environ Med. 2008 Jun;79(6):585-90. doi: 10.3357/asem.2245.2008. PMID 18581942
- [Background] Spalding JA, Cole BL, Mir FA. Advice for medical students and practitioners with colour vision deficiency: a website resource. Clin Exp Optom. 2010 Jan;93(1):39-41. doi: 10.1111/j.1444-0938.2009.00434.x. Epub 2009 Oct 27. No abstract available. PMID 19863590
- [Background] Rabin J. Cone-specific measures of human color vision. Invest Ophthalmol Vis Sci. 1996 Dec;37(13):2771-4. PMID 8977494
- [Background] Rabin J. Quantification of color vision with cone contrast sensitivity. Vis Neurosci. 2004 May-Jun;21(3):483-5. doi: 10.1017/s0952523804213128. PMID 15518234
- [Background] Rabin J, Gooch J, Ivan D. Rapid quantification of color vision: the cone contrast test. Invest Ophthalmol Vis Sci. 2011 Feb 9;52(2):816-20. doi: 10.1167/iovs.10-6283. PMID 21051721
- [Background] Werner JS, Marsh-Armstrong B, Knoblauch K. Adaptive Changes in Color Vision from Long-Term Filter Usage in Anomalous but Not Normal Trichromacy. Curr Biol. 2020 Aug 3;30(15):3011-3015.e4. doi: 10.1016/j.cub.2020.05.054. Epub 2020 Jun 25. PMID 32589909
- [Background] Rabin JC, Kryder AC, Lam D. Diagnosis of Normal and Abnormal Color Vision with Cone-Specific VEPs. Transl Vis Sci Technol. 2016 May 17;5(3):8. doi: 10.1167/tvst.5.3.8. eCollection 2016 May. PMID 27226932
- [Background] Rabin J, Kryder A, Lam D. Binocular facilitation of cone-specific visual evoked potentials in colour deficiency. Clin Exp Optom. 2018 Jan;101(1):69-72. doi: 10.1111/cxo.12567. Epub 2017 Jun 21. PMID 28636141
- [Background] Rabin J, Silva F, Trevino N, Gillentine H, Li L, Inclan L, Anderson G, Lee E, Vo H. Performance enhancement in color deficiency with color-correcting lenses. Eye (Lond). 2022 Jul;36(7):1502-1503. doi: 10.1038/s41433-021-01924-0. Epub 2022 Jan 8. No abstract available. PMID 34999724

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT05463016/Prot_SAP_ICF_000.pdf